CLINICAL TRIAL: NCT01947946
Title: A Multicentre, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase III Efficacy and Safety Study of Benralizumab (MEDI-563) Added to Medium-dose Inhaled Corticosteroid Plus Long-acting β2 Agonist in Patients With Uncontrolled Asthma
Brief Title: Efficacy and Safety Study of Benralizumab Added to Medium-dose Inhaled Corticosteroid Plus LABA in Patients With Uncontrolled Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to sponsor decision
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00016
Record Dates: First submitted 2013-09-11; First posted 2013-09-23 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benra 30 mg q.4 Weeks (Experimental): Fixed 30 mg dose of benralizumab (every 4 weeks)
  Interventions: Biological: Benralizumab
- Benra 30 mg - Placebo q.8 Weeks (Experimental): Fixed 30 mg dose of benralizumab, every 4 weeks for the first 3 doses and then every 8 weeks thereafter, (placebo injections administered at the 4 week interim treatment visits to maintain blind).
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): A (Dummy) injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benra 30 mg q.4 Weeks is a fixed 30 mg dose of benralizumab subcutaneously on study week 0 until study week 44 inclusive.
  Benra 30 mg - Placebo q.8 Weeks is a fixed 30 mg dose of benralizumab, every 4 weeks for the first 3 doses and then every 8 weeks thereafter, (placebo injections administrated at the 4 week interim visits to maintain blind). It is subcutaneously administered on study week 0 until study week 44 inclusive.
  Arms: Benra 30 mg - Placebo q.8 Weeks; Benra 30 mg q.4 Weeks
Biological: Placebo — Placebo subcutaneously on study week 0 until study week 44 inclusive.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Benralizumab reduces the number of asthma exacerbations in patients who remain uncontrolled on medium doses of ICS-LABA.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and male aged from 18 to 75 years, inclusively
3. History of physician-diagnosed asthma requiring treatment with medium dose ICS (>250ug fluticasone dry powder formulation equivalents total daily dose) and a LABA, for at least 12 months prior to Visit 1
4. Documented treatment with medium-dose ICS (>250ug and ≤500ug fluticasone dry powder formulation equivalents total daily dose) and LABA for at least 3 month prior to Visit 1

Exclusion criteria:

1. Clinically important pulmonary disease other than asthma (e.g. active lung infection, COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg- Strauss syndrome, hypereosinophilic syndrome)
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could: - Affect the safety of the patient throughout the study - Influence the findings of the studies or their interpretations - Impede the patient's ability to complete the entire duration of study
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period 4. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening/run-in period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W. Busse, MD, Principal Investigator — Allergy, Pulmonary and Critical Care Medicine, Clinical Science Center 600 Highland Ave, Madison, WI USA
Locations (47):
- United States (21):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, San Jose, California
  - Research Site, Centennial, Colorado
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Rock Hill, South Carolina
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugarland, Texas
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aire
- Research Site, São Paulo, Brazil
- Bulgaria (3):
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Germany (2):
  - Research Site, Hamburg
  - Research Site, Mainz
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Giżycko
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żnin
- Russia (10):
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Ulyanovsk
  - Research Site, Vladikavkaz
  - Research Site, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was stopped with 13 patients randomised
Groups:
- Benra 30 mg q.4 Weeks: Fixed 30 mg dose of benralizumab every 4 weeks.
- Benra 30 Mg-Placebo q.8 Weeks: Fixed 30 mg dose of benralizumab, every 4 weeks for the first 3 doses and then every 8 weeks thereafter, (placebo injections administered at the 4 week interim treatment visits to maintain blind).
Period: Overall Study
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 Mg-Placebo q.8 Weeks | Placebo
Started | 3 | 5 | 5
Completed | 0 (Study Stopped) | 0 | 0
Not Completed | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis will be from the full analysis set. The full analysis set consists of all patients randomized and receiving any investigational product, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 Mg-Placebo q.8 Weeks | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (15.70) | 57.8 (6.38) | 49.6 (6.35) | 54.8 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Asthma Exacerbations Over 48 Weeks Treatment
Description: The number of asthma exacerbations over 48 weeks treatment will be counted
Time Frame: 48 weeks treatment
Population: Patients from the full analysis set will be used. All patients randomized and receiving any investigational product will be included in the full analysis set, irrespective of their protocol adherence and continued participation in the study.
Measure: Number; unit: Number of events
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 Mg-Placebo q.8 Weeks | Placebo
Number analyzed (Participants) | 3 | 3 | 3
Number of events | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 Mg-Placebo q.8 Weeks | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg q.4 Weeks (N=3) | Benra 30 Mg-Placebo q.8 Weeks (N=5) | Placebo (N=5)
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No